CLINICAL TRIAL: NCT00968383
Title: Late Percutaneous Coronary Intervention of the Occluded Infarct-Related Artery in Patients With Preserved Infarct Zone Viability Determined With Magnetic Resonance Imaging
Brief Title: Cardiovascular Magnetic Resonance for the Occluded Infarct-Related Artery Treatment
Acronym: COAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely terminated due to low enrollment.
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.50/V/09
Record Dates: First submitted 2009-06-30; First posted 2009-08-31 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Heart Failure
Keywords: Acute Coronary Syndrome; Myocardial infarction; Infarct Related Artery; Percutaneous Coronary Intervention; Medical treatment; Tissue Viability; Magnetic Resonance
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Heart Failure; Acute Coronary Syndrome | interventions — Adrenergic beta-Antagonists; Platelet Aggregation Inhibitors; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimal medical therapy (Active Comparator): Conventional medical management, including aspirin, clopidogrel, statins, beta blockers, angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blocker (ARB) and/or aldosterone antagonist and risk factor modification
  Interventions: Drug: Beta adrenergic blockers; Drug: Platelet inhibitors; Drug: Statins; Drug: ACE inhibitors and/or ARB and/or AA
- PCI with optimal medical therapy (Experimental): Conventional medical management, including aspirin, clopidogrel, statins, beta blockers, angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blocker (ARB) and/or aldosterone antagonist and risk factor modification plus percutaneous coronary intervention and coronary stenting
  Interventions: Drug: Beta adrenergic blockers; Drug: Platelet inhibitors; Drug: Statins; Drug: ACE inhibitors and/or ARB and/or AA; Procedure: PCI with stenting

INTERVENTIONS:
Drug: Beta adrenergic blockers — Participants will receive beta adrenergic blockers.
Drug: Platelet inhibitors — Participants will receive platelet inhibitors.
Drug: Statins — Participants will receive statins.
Drug: ACE inhibitors and/or ARB and/or AA — Participants will receive ACE inhibitors and/or ARB and/or AA
Procedure: PCI with stenting — Participants will undergo percutaneous coronary intervention (PCI) and coronary stenting.
  Arms: PCI with optimal medical therapy

SUMMARY:
The purpose of this study is to determine whether opening an occluded infarcted artery 3-28 days after an acute myocardial infarction in high-risk asymptomatic patients with preserved infarct zone viability improves left ventricular systolic function and volumes at 6 months follow-up. The secondary purpose is to assess the changes in myocardial tissue characteristics after late percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Rapid restoration of blood flow in the infarct-related artery (IRA), one of the cornerstones of contemporary treatment of acute myocardial infarction (MI) prevents myocardial necrosis and its consequences. However, due to late presentation or failed fibrinolytic therapy up to one third of patients have persistently occluded IRA after MI.

Recently, the Occluded Artery Trial (OAT) has demonstrated that percutaneous coronary intervention (PCI) with optimal medical therapy does not reduce the frequency of major adverse events compared to optimal medical therapy alone when performed on days 3-28 post MI in stable patients. Assessment of infarct zone viability was not used as an inclusion/exclusion criterion in the main OAT trial.

Several studies confirm that patients with left ventricular systolic dysfunction and preserved myocardial viability (necrosis transmurality<50% in most segments of the infarct zone) assessed with magnetic resonance imaging benefit from revascularization.

Late opening of the occluded infarct-related artery only in patients with preserved myocardial tissue viability may lead to improvement of left ventricular volumes and function.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment 3-28 days after an acute myocardial infarction.
* Infarct related artery occlusion (TIMI 0 or 1).
* High risk: left ventricular ejection fraction (LVEF)<50% or LVEF>50% and proximal coronary occlusion.
* Preserved infarct zone viability (necrosis transmurality <50% in at least 4 segments out of 17 according to AHA classification).

Exclusion Criteria:

* Unstable clinical condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
change in systolic wall thickening (SWT) | 6 months

SECONDARY OUTCOMES:
change in left ventricular ejection fraction (LVEF) | 6 months
change in wall motion score index (WMSI) | 6 months
change in left ventricular end-diastolic volume (LVEDV) | 6 months
change in left ventricular end-systolic volume (LVESV) | 6 months
myocardial tissue characteristics | 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz A Malek, M.D. PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Mariusz Kruk, M.D. PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland; Mariusz Klopotowski, M.D., Study Chair — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Background] Hochman JS, Lamas GA, Knatterud GL, Buller CE, Dzavik V, Mark DB, Reynolds HR, White HD; Occluded Artery Trial Research Group. Design and methodology of the Occluded Artery Trial (OAT). Am Heart J. 2005 Oct;150(4):627-42. doi: 10.1016/j.ahj.2005.07.002. PMID 16209957
- [Background] Hochman JS, Lamas GA, Buller CE, Dzavik V, Reynolds HR, Abramsky SJ, Forman S, Ruzyllo W, Maggioni AP, White H, Sadowski Z, Carvalho AC, Rankin JM, Renkin JP, Steg PG, Mascette AM, Sopko G, Pfisterer ME, Leor J, Fridrich V, Mark DB, Knatterud GL; Occluded Artery Trial Investigators. Coronary intervention for persistent occlusion after myocardial infarction. N Engl J Med. 2006 Dec 7;355(23):2395-407. doi: 10.1056/NEJMoa066139. Epub 2006 Nov 14. PMID 17105759
- [Background] Malek LA, Reynolds HR, Forman SA, Vozzi C, Mancini GB, French JK, Dziarmaga M, Renkin JP, Kochman J, Lamas GA, Hochman JS. Late coronary intervention for totally occluded left anterior descending coronary arteries in stable patients after myocardial infarction: Results from the Occluded Artery Trial (OAT). Am Heart J. 2009 Apr;157(4):724-32. doi: 10.1016/j.ahj.2008.12.008. PMID 19332202
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Derived] Malek LA, Silva JC, Bellenger NG, Nicolau JC, Klopotowski M, Spiewak M, Rassi CH, Lewandowski Z, Kruk M, Rochitte CE, Ruzyllo W, Witkowski A. Late percutaneous coronary intervention for an occluded infarct-related artery in patients with preserved infarct zone viability: a pooled analysis of cardiovascular magnetic resonance studies. Cardiol J. 2013;20(5):552-9. doi: 10.5603/CJ.2013.0141. PMID 24297771